CLINICAL TRIAL: NCT01562626
Title: A Phase I/II Safety, Pharmacokinetic, and Pharmacodynamic Study of APS001F With Flucytosine and Maltose for the Treatment of Advanced and/or Metastatic Solid Tumors
Brief Title: Phase I/II Study of APS001F With Flucytosine and Maltose in Solid Tumors
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anaeropharma Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APS001F-001
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Tumors; Neoplasms; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Flucytosine; Maltose

ARMS (1):
- Dose escalation (Experimental)
  Interventions: Drug: APS001F; Drug: Flucytosine (5-FC); Drug: 10% maltose

INTERVENTIONS:
Drug: APS001F — APS001F infusion on Days 1,2,3 of each 28 day cycle.
Drug: Flucytosine (5-FC) — oral doses on Days 11-15 and 18-22, each 28 day cycle
Drug: 10% maltose — 10% maltose infusion will be administered on Days 1-5, 8-12, and 15-19, each 28 day cycle.

SUMMARY:
The purpose of this study is to test the safety and efficacy of an investigational drug called APS001F when given with flucytosine (5-FC) for treatment of solid tumors. APS001F is a recombinant Bifidobacterium longum (a live bacteria normally found in the digestive tract) that has been modified to produce an enzyme, cytosine deaminase (CD). The patient will first receive an injection of APS001F followed by oral 5-FC. APS001F is expected to go to the site of the tumor(s) where the agent will produce CD enzyme. CD enzyme will convert the 5-FC into 5-fluorouracil (5-FU) which is a standard chemotherapy drug for several types of cancer. Additionally, some patients will also receive 10% maltose injection, a sugar that has been shown to enhance the growth and effectiveness of APS001F in animals. This is the first study where APS001F is being used in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced and/or metastatic, histologically documented solid tumors.
2. Patients must have disease that is no longer considered responsive to available conventional modalities or treatments (failed any known standard curative or effective therapy for that disease).
3. Patients must have measurable or evaluable advanced and/or metastatic disease by RECIST 1.1.
4. Patients enrolled at Dose Level 6 or higher in the phase I portion of the trial must have at least one tumor mass suitable and easily accessible for excisional biopsy, or alternatively, accessible for CT or ultrasound guided core needle biopsy. The procedure must be able to be performed with minimum morbidity.
5. ECOG Performance status of 0 or 1.
6. Must be at least 18 years of age.
7. Expected survival of at least 3 months.
8. Men and women of child-bearing potential (i.e., women who are premenopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device (IUD), oral contraceptive or double barrier device), and women must have a negative serum or urine pregnancy test 1 week before beginning treatment on this trial. Nursing patients are also excluded.
9. Must be able and willing to give written informed consent.
10. Patients must have adequate major organ function and meet the following criteria:

    * white blood cell (WBC)count >= 3,000/mm3.
    * Absolute neutrophil count (ANC) >= 1500/uL.
    * Platelets >= 100,000/mm3.
    * Hemoglobin >= 9.0g/dL
    * Serum creatinine <= 1.5 mg/dL. (or estimated creatinine clearance >= 50 ml/min/1.73 m2)
    * Bilirubin <= 1.5 mg/dL; ALT, AST, and alkaline phosphatase <= 3.0x the upper limit of normal
    * Prothrombin Time (PT) and activated partial thromboplastin time (aPTT) <= 1.5x the upper limit of normal.
    * Oxygen saturation >= 90% by pulse oximetry
11. Patients should have body Temperature <= 38.0 degrees C.
12. Echocardiogram demonstrated left ventricular ejection fraction >= 40%.

Exclusion Criteria:

1. Presence or history of brain metastases.
2. Presence of known or suspected ongoing ischemia of non-tumor tissues including

   * ischemic peripheral vascular disease, myocardial infarction within the past 6 months,
   * congestive heart failure > class II NYHA,
   * unstable angina (anginal symptoms at rest) or new onset angina (i.e., began within the last 3 months).
   * cerebrovascular accident, including transient ischemic attacks within the past 6 months.
3. An artificial implant that cannot be easily removed (e.g., heart valves, prosthetic hips or knees, or other devices), which could allow a nidus of infection.
4. Patients with indwelling catheters (other than Portacath, Hickman or PICC lines)
5. Known cardiac valvular disease (e.g. bicuspid aortic valve) or arterial aneurysm(s) that may allow a nidus of infection.
6. Known cardiac arrhythmias requiring medication.
7. Patients with any of the following cardiovascular conditions: patent foramen ovale, prior history of bacterial endocarditis, any existing thrombus (either arterial or venous) as well as known history of DVT, permanent pacemakers, AICDs, LVADs, or other intravascular cardiac device, known AV malformations.
8. Patients with baseline respiratory insufficiency severe enough to require supplemental oxygen.
9. Patients with pleural effusion or abdominal/peritoneal ascites, except the finding of physiological levels of fluid.
10. Patients who have not fully recovered from toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment). The required minimum time elapsed from prior treatments are:

    * treatment with cytotoxic agents, or treatment with biologic agents within 4 weeks prior to treatment with APS001F (6 weeks for mitomycin C or nitrosoureas).
    * treatment with molecular targeted agents within 2 weeks prior to treatment with APS001F.
    * radiotherapy within 4 weeks prior to treatment with APS001F (intensive radiotherapy within 6 weeks or palliative radiotherapy within 2 weeks).
    * At least 2 weeks must have elapsed from any prior surgery or hormonal therapy.
11. Presence of GI bleeding.
12. Currently using warfarin.
13. Active infection of any kind.
14. Currently using antibiotics and/or anti fungal agent (however, topical antibiotics are permitted).
15. Presence of any condition or concurrent requirement for treatment with agents known to result in immune deficiency.
16. Patients with documented immunodeficiency such as HIV infection.
17. Presence of autoimmune disease that requires corticosteroids and/or immunosuppressive agents.
18. Patients with evidence of chronic active Hepatitis B (positive for HbsAg) and Hepatitis C (positive for viral RNA).
19. Hypersensitivity (history of allergic reactions) to

    * 5-FC
    * 5-FU
20. Patient's medical history does not contraindicate treatment with at least one of the following antibiotics: ampicillin, clindamycin and erythromycin/clarithromycin.
21. Unwilling or unable to follow protocol requirements.
22. Presence of any concurrent illness or condition that, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-09; Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of APS001F treatment plus 5-FC and maltose | Starting from date of first dose up to 30 days after last dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - MD Anderson, Houston, Texas